CLINICAL TRIAL: NCT04542759
Title: Effect of Topical Besifloxacin on Ocular Surface Bacterial Microbiota Prior to Cataract Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI-004-215
Record Dates: First submitted 2020-08-19; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Microbial Disease; Cataract Senile
Keywords: Besifloxacin; prophylaxis; cataract surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Besifloxacin (Active Comparator): 1 DROP 4 TIMES A DAY FOR 3 DAYS PRIOR SURGERY
  Interventions: Drug: Besifloxacin Ophthalmic
- Hydroxypropyl methylcellulose (Placebo Comparator): 1 DROP 4 TIMES A DAY FOR 3 DAYS PRIOR SURGERY
  Interventions: Drug: Hydroxypropyl Methylcellulose Ophthalmic Ophthalmic Solution

INTERVENTIONS:
Drug: Besifloxacin Ophthalmic — Prophylaxis for endophthalmitis
  Other Names: Besivance ophthalmic suspension 0.6%
  Arms: Besifloxacin
Drug: Hydroxypropyl Methylcellulose Ophthalmic Ophthalmic Solution — Placebo
  Other Names: Artelac eye drops
  Arms: Hydroxypropyl methylcellulose

SUMMARY:
Describe the efficacy of the use of topical besifloxacin in reducing the conjunctival microbiota as a prophylactic measure in patients scheduled for cataract surgery.

DETAILED DESCRIPTION:
Randomized double-blind clinical trial. Study carried out in a single center between January and April 2017. 60 eyes were included that were randomly divided in a 1: 1 ratio into two groups. The first group received placebo (hydroxypropylmethylcellulose drops) while the second group received 0.6% besifloxacin drops four times a day for 3 days. All of them had a conjunctival cul-de-sac culture before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age scheduled for cataract surgery in the established study period.
* Subjects physically and mentally capable of applying the eye drops or having a person available to help in the correct administration of the eye drops 4 times a day.

Exclusion Criteria:

* - Active eye infection (bacterial, viral, fungal or parasitic) such as blepharitis and / or conjunctivitis.
* Known allergy or any contraindication to the use of quinolones or any of the components of the drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Percentage of positive cultures before and after treatment in each arm | Through study completion, an average of 1 year
  A conjunctival cul-de-sac sample will be taken before starting treatment and before surgery, which will be cultured on 3 different media types: Blood, Chocolate and Sabouraud agar.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Chavez-Mondragon, MD, Study Director — Instutute of Ophthalmology "Conde de Valenciana"
Locations (1):
- Institute of Ophthalmology, Conde de Valenciana Foundation, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No